CLINICAL TRIAL: NCT00711295
Title: An Open-Label Phase 3 Study to Assess the Safety and Immunogenicity of a Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine in an Adult and Elderly Population as Well as in Specified Risk Groups
Brief Title: Phase 3 Study of a H5N1 Vaccine in Adults, Elderly and Specified Risk Groups
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Yuri Martina PhD (Clinical Project Manager), Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 810705
Record Dates: First submitted 2008-07-02; First posted 2008-07-08 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2010-11

CONDITIONS: Influenza
Keywords: Influenza (Pandemic)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1, Treatment Arm 1 (Experimental): Stratum A (18-59 ys)/B(>=60 ys): 120 healthy volunteers per stratum will receive 2 vaccinations with 7.5 µg A/Vietnam/1203/2004 on Days 0 and 21 and participate in immunogenicity evaluation.
  Among Stratum A volunteers, 60 will participate in antibody kinetics evaluation and 30 in cellular immunity evaluation.
  Randomization to Treatment Arms 1 and 2 at 2:1 ratio. Subjects in Treatment Arm 1 will be included in the immunologic determination of lot-to-lot consistency.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted
- Cohort 1, Treatment Arm 2 (Experimental): Stratum A (18-59 ys)/B(>=60 ys): 60 healthy volunteers per stratum will receive 2 vaccinations with 3.75 µg A/Vietnam/1203/2004 on Days 0 and 21 and participate in immunogenicity evaluation.
  Randomization to Treatment Arms 1 and 2 at 2:1 ratio.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted
- Cohort 1, Treatment Arm 3 (Experimental): Stratum A (18-59 ys): 2060 healthy volunteers will receive 2 vaccinations with 7.5 µg A/Vietnam/1203/2004 on Days 0 and 21 and participate in safety evaluation only.
  Randomization within Treatment Arms 3 and 4 at 1:1:1 ratio per study site to receive one of three different lots of the H5N1 influenza vaccine.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted
- Cohort 2, Treatment Arm 1 (Experimental): 300 immune compromised individuals 18 years or older will receive 2 vaccinations with 7.5 µg A/Vietnam/1203/2004 on Days 0 and 21.
  100 will participate in immunogenicity evaluation and 30 in cellular immunity evaluation.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted
- Cohort 3, Treatment Arm 1 (Experimental): 300 chronically ill patients 18 years or older will receive 2 vaccinations with 7.5 µg A/Vietnam/1203/2004 on Days 0 and 21 and participate in immunogenicity evaluation.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted
- Cohort 1, Treatment Arm 4 (Experimental): Stratum A (18-59): 540 healthy volunteers will receive 2 vaccinations with 7.5 µg A/Vietnam/1203/2004 on Days 0 and 21 and participate in immunogenicity assessment.
  Randomization within Treatment Arms 3 and 4 at 1:1:1 ratio per study site to receive one of three different lots of the H5N1 influenza vaccine.
  Subjects in Treatment Arm 4 will be included in the immunologic determination of lot-to-lot consistency.
  Interventions: Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted

INTERVENTIONS:
Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted — Intramuscular injection of 7.5 µg hemagglutinin antigen (A/Vietnam/1203/2004 strain) in a non-adjuvanted formulation on Days 0 and 21.
  Arms: Cohort 1, Treatment Arm 1; Cohort 1, Treatment Arm 3; Cohort 1, Treatment Arm 4; Cohort 2, Treatment Arm 1; Cohort 3, Treatment Arm 1
Biological: H5N1 Influenza Vaccine Whole virion, Vero cell-derived, Inactivated Influenza Vaccine, non-adjuvanted — Intramuscular injection of 3.75 µg hemagglutinin antigen (A/Vietnam/1203/2004 strain) in a non-adjuvanted formulation on Days 0 and 21.
  Arms: Cohort 1, Treatment Arm 2

SUMMARY:
The purpose of this study is to assess the safety and tolerability of, and the immune response to a non-adjuvanted H5N1 influenza vaccine in an adult and elderly population and in specified risk groups. Furthermore, persistence of H5N1 influenza antibodies after vaccination with this vaccine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria apply to subjects in all three cohorts:

Male and female subjects will be eligible for participation in this study if they:

* Are 18 years of age or older on the day of screening;
* Have an understanding of the study and its procedures, agree to its provisions, and give written informed consent prior to study entry;
* Are physically and mentally capable of participating in the study and follow its procedures;
* Agree to keep a daily record of symptoms for the duration of the study;
* If female of childbearing potential - have a negative urine pregnancy test result within 24 hours prior to the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study.

The following inclusion criterion applies to subjects in Cohort 1 only:

- Are generally healthy [1], as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination.

([1]) Subjects with controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90-99 mmHg diastolic) are eligible for participation in Cohort 1 of this study.

The following inclusion criterion applies to subjects in Cohort 2 only:

- Are immune compromised due to immunosuppressive treatment (e.g. transplant patients [2]) or due to acquired immunodeficiency caused by HIV infection with or without treatment with anti-retrovirals.

([2]) Transplant patients should be at least 6 months after transplantation and in stable clinical condition without complications.

The following inclusion criterion applies to subjects in Cohort 3 only:

- Have a chronic cardiovascular (excluding hypertension) [3], respiratory, renal, or metabolic (e.g. diabetes mellitus) illness in stable clinical condition without major disease complications such as organ failure, infectious complications, severe asthma or respiratory dysfunction.

([3]) Subjects with cardiovascular disease such as coronary heart disease, angina, heart attack or other heart conditions in stable clinical condition, without major disease complications and who are considered at risk for medical complications from influenza. However, subjects with hypertension (see [1] above) not associated with any heart condition will be excluded from participation in Cohort 3 of this study.

Exclusion Criteria:

The following exclusion criteria apply to subjects in all three cohorts:

Subjects will be excluded from participation in this study if they:

* Have a history of exposure to H5N1 virus or a history of vaccination with an H5N1 influenza vaccine;
* Are at high risk of contracting H5N1 influenza infection (e.g. poultry workers);
* Have a history of severe allergic reactions or anaphylaxis;
* Have a rash, dermatological condition or tattoos which may interfere with injection site reaction rating;
* Have donated blood or plasma within 30 days prior to study entry;
* Have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study;
* Have a known or suspected problem with alcohol or drug abuse;
* Were administered an investigational drug within 6 weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product;
* Are a member of the team conducting this study or are in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study;
* If female: are pregnant or lactating.

The following exclusion criteria apply to subjects in Cohort 1 only:

* Currently have or have a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder [4];
* Have any inherited or acquired immunodeficiency;
* Have a disease or are currently undergoing a form of treatment or were undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs;
* Have received a blood transfusion or immunoglobulins within 90 days prior to study entry;
* Have a functional or surgical asplenia.

([4]) A significant disorder is defined as a disease or medical condition associated with impaired health status, increased risk for complications, requiring medical treatment and/or follow up.

The following exclusion criteria apply to subjects in Cohort 2 only:

* Are immune compromised due to stem cell or organ-transplantation with significant medical complications such as acute or chronic graft rejection or graft versus host disease requiring intensive immunosuppressive treatment, transplant failure or infectious complications or other conditions that would be considered a contraindication for vaccination with an inactivated vaccine.
* Are immune compromised due to HIV infection with a CD4 count of < 200x10^6/L at screening or significant medical complications such as opportunistic infections, malignant complications (e.g. lymphoma, Kaposi sarcoma), other organ manifestations consistent with advanced acquired immunodeficiency syndrome (AIDS) or other conditions that would be considered a contraindication for vaccination with an inactivated vaccine.

The following exclusion criterion applies to subjects in Cohort 3 only:

- Have a chronic cardiovascular, respiratory, renal, or metabolic (e.g. diabetes mellitus) illness with significant complications such as advanced heart failure, liver failure, renal failure, severe asthma or severe respiratory failure, infectious complications or other conditions that would be considered a contraindication for vaccination with an inactivated vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3583 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of systemic reactions until 21 days after the first and second vaccinations | 42 days
Number of subjects with antibody response to the vaccine strain associated with protection 21 days after the second vaccination defined as titer measured by microneutralization (MN) assay >= 1:20. | 42 days
Antibody response 21 days after the second vaccination as measured by MN assay; | 42 days

SECONDARY OUTCOMES:
Frequency and severity of injection site reactions until 21 days after the first and second vaccinations | 42 days
Number of subjects with fever, malaise or shivering with onset within 7 days after the first and second vaccinations | 7 days
Frequency and severity of adverse events observed during the entire study period | 11 months
Number of subjects with antibody response associated with protection 21 days after the first and second vaccinations defined as Hemagglutination Inhibition Antibody (HIA) titer >= 1:40 or Single Radial Hemolysis (SRH) area >= 25 mm2 | 42 days
Number of subjects with antibody response associated with protection 21 days after the second vaccination defined as titer measured by MN assay >=1:40, >= 1:80, >=1:160 | 42 days
Antibody response 21 days after the first and second vaccinations as measured by HI and SRH assays | 42 days
Fold increase of antibody response 21 days after the first and second vaccinations as compared to baseline as measured by MN, HI and SRH assays | 42 days
Number of subjects with seroconversion (MN/HI: min.4-fold titer increase vs baseline;SRH:post-vacc. hemolysis area >=25mm2 or increased by >=50% for pre-vacc. sample <=4mm2 and >4mm2, resp., 21 days after 1st and 2nd vaccinations, measured by MN,HI,SRH | 42 days
Number of subjects with antibody response associated with protection 201 days after the first vaccination as measured by MN, HI and SRH assays | 201 days
Antibody response 201 days after the first vaccination as measured by MN, HI and SRH assays | 201 days
Fold increase of antibody response 201 days after the first vaccination as compared to baseline as measured by MN, HI and SRH assays | 201 days
Number of subjects in the subset included in the assessment of antibody kinetics with antibody response associated with protection 28, 35 and 90 days after the first vaccination as measured by MN, HI and SRH assays | 90 days
Antibody response in the subset of subjects included in the assessment of antibody kinetics 28, 35 and 90 days after the first vaccination as measured by MN, HI and SRH assays | 90 days
Fold increase of antibody response in the subset of subjects included in the assessment of antibody kinetics 28, 35 and 90 days after the first vaccination as compared to baseline as measured by MN, HI and SRH assays | 90 days
Number of subjects in subset for antibody kinetics evaluation with seroconversion (see definitions above) 28, 35, 90 days after 1st vaccination, measured by MN, HI, SRH | 90 days
T-cell response in the subset of subjects included in the evaluation of cellular immunity after each vaccination as determined by the frequency of cytokine producing T-cells induced by influenza virus antigens | 201 days
Increase in frequency of cytokine producing T-cells induced by influenza virus antigens after each vaccination as compared to baseline | 201 days
Number of subjects with antibody response associated with protection 21 days after the first vaccination defined as titer measured by MN assay >=1:20, >=1:40, >=1:80, >=1:160 | 21 days
Antibody response 21 days after the first vaccination as measured by MN assay | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Bio Science Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (45):
- Austria (3):
  - Allgemeines Krankenhaus Wien, Innere Medizin, Waehringer Guertel 18-20, Vienna
  - Institut für spezifische Prophylaxe und Tropenmedizin, Kinderspitalgasse 15, Vienna
  - University Clinic for Clinical Pharmacology, Vienna Medical University / Vienna General Hospital, Waehringer Guertel 18-20, Vienna
- Belgium (5):
  - OLV Hospital Aalst, Research Unit, Moorselbaan 164, Aalst
  - Cliniques Universitaires Saint Luc, Avenue Hippocrate 10, Niveau -1 Couloir C11, Brussels
  - Center for Vaccinologie, UZ Gent, De Pintelaan 185, Ghent
  - UZ Leuven, Kapucijnenvoer 35, Block D, Box 7001, Leuven
  - UZ Antwerpen, Universiteitsplein 1, Wilrijk
- Finland (5):
  - Espoon rokotetutkimusklinikka, Keskustorni 7. krs., Tapiontori 1, Espoo
  - Etelä-Helsingin rokotetutkimusklinikka, Vuorikatu 18, 3 krs, Helsinki
  - Tampereen rokotetutkimusklinikka, Pinninkatu 47, 1.krs, Tampere
  - Turun rokotetutkimusklinikka, Lemminkäisenkatu 14-18 B, 4.krs, Turku
  - Itä-Vantaan rokotetutkimusklinikka, Asematie 11 A 16, Vantaa
- Germany (11):
  - Charité - Universitaetsmedizin Berlin, Medizinische Klinik III, Haematologie, Onkologie & Transfusionsmedizin, Karl Landsteiner-Haus, 1 OG, Hindenburgdamm 30, Berlin
  - Klinische Forschung Berlin Buch GmbH, Robert-Rössle-Str. 10 / Haus 85, Berlin
  - Klinikum der Universitaet zu Koeln, Klinik I für Innere Medizin, Studienbüro für Infektiologie, Haus 11, Kerpener Str. 62, Cologne
  - Carl Gustav Carus Universitaet, Medizinische Klinik und Poliklinik I, Haematologie/Onkologie Fetscherstr. 74, Dresden
  - Klinikum der J.W.Goethe Universitaet, Medizinische Klinik II Schwerpunkt HIV Haus 68, Theodor-Stern-Kai 7, Frankfurt am Main
  - Klinische Forschung Hamburg GmbH, Hoheluftchaussee 18, Hamburg
  - Universitätsklinikum Leipzig, Selbstständige Abteilung für Hämatologie, Internistische Onkologie und Hämostaseologie, Johannisallee 32A, Leipzig
  - Johannes Gutenberg Universitaet, I. Medizinische Klinik und Poliklinik, Langenbeckstr. 1, Mainz
  - Johannes Gutenberg-Universitaet, III. Medizinische Klinik und Poliklinik, Langenbeckstr. 1, Mainz
  - Studienzentrum Mainz-Mitte am GesundheitsCentrum Mainz, Große Langgasse 1A/Eingang Kötherhofstrasse 4, Mainz
  - Institut für Tropenmedizin, Wilhelmstraße 27, Tübingen
- Latvia (7):
  - Private practice, Berzpils street 14-16, Balvi
  - Outpatient clinic " Jelgavas centra doktorats ", Kr. Barona str. 17, Jelgava
  - Private practice, Aptiekas maja, Madliena village, Ogres district, Madlienas Parish
  - Outpatient clinic "Alma", Kr.Valdemara street 20-4, Riga
  - Outpatient clinic "Adoria", Caka street 70-3, Riga
  - Outpatient clinic "Veselibas centrs-4", Kr.Barona str. 117, Riga
  - Private practice, Slimnicas street 3, Saldus
- Lithuania (7):
  - Kaunas 2nd Clinical Hospital, Clinic of Infectious Diseases, Baltijos ave. 120, Kaunas
  - Silainiai Family Health Center, Baltu ave. 7a, Kaunas
  - Saules Family Medicine Center, Birzelio 23 ios. 4, Kaunas
  - Klaipeda University Hospital, Department of Infectious Diseases, Liepojos str. 41, Klaipėda
  - Institute of Psychophysiology and Rehabilitation of Kaunas University of Medicine, Vyduno 4, Palanga
  - Siauliai District Hospital, Infectious Diseases, Kudirkos 99, Šiauliai
  - National Tuberculosis and Infectious Diseases University Hospital, Vilnius University Clinic of Infectious Diseases, Dermatovenereology and Microbiology, Birutes street 1/20, Vilnius
- Netherlands (7):
  - Andromed Breda, Middellaan 5, Breda
  - Andromed Eindhoven B.V., Bomanshof 6, Eindhoven
  - Andromed Noord B.V., Damsterdiep 9, Groningen
  - Andromed Leiden B.V., Doezastraat 1 GZ, Leiden
  - Andromed, Kamerlingh Onnestraat 16 -18, Nijmegen
  - Andromed Oost B.V., Reigerstraat 30E, Velp
  - Andromed Zoetermeer, Parkdreef 142, Zoetermeer

REFERENCES:
- [Derived] van der Velden MV, Geisberger A, Dvorak T, Portsmouth D, Fritz R, Crowe BA, Herr W, Distler E, Wagner EM, Zeitlinger M, Sauermann R, Stephan C, Ehrlich HJ, Barrett PN, Aichinger G. Safety and immunogenicity of a vero cell culture-derived whole-virus H5N1 influenza vaccine in chronically ill and immunocompromised patients. Clin Vaccine Immunol. 2014 Jun;21(6):867-76. doi: 10.1128/CVI.00065-14. Epub 2014 Apr 16. PMID 24739978